CLINICAL TRIAL: NCT03995186
Title: Effects of Behavioural Activation on Emotional Cognition and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Principal Investigator, Catherine Harmer, Professor, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Beh_Act_ETB
Record Dates: First submitted 2019-04-23; First posted 2019-06-21 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Depression; Depressive Disorder; Mood Disorders; Cognition
Keywords: behavioural activation
MeSH Terms: conditions — Depression; Depressive Disorder; Mood Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the behavioural activation intervention (40 participants), activity monitoring (40 participants) or passive waiting-list control group (40 participants). This study is not intended to be administering treatment, it is investigating the possible mechanisms of this intervention.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Behavioural activation group (Experimental)
  Interventions: Behavioral: Behavioural activation
- Activity monitoring group (Active Comparator)
  Interventions: Behavioral: Activity monitoring
- Waiting list control group (No Intervention)

INTERVENTIONS:
Behavioral: Behavioural activation — 4-week programme based on the behavioural activation treatment provided in the NHS IAPT services. The programme includes psychoeducation on the relationship between activity and depression, examining the depressed person's level of activity, helping them identify activities they would like to increase and supporting them in the planning and conduct of those activities.
  Arms: Behavioural activation group
Behavioral: Activity monitoring — 4-week programme where participants simply monitor their general daily activities in a diary.
  Arms: Activity monitoring group

SUMMARY:
Behavioural activation (BA) is widely accepted as an efficacious treatment for depression. It has been suggested that several depression treatments work via early changes in emotional processing (e.g. affective bias in the processing of facial expressions) and that these could help predict treatment success, but it has not yet been examined whether the same applies in behavioural interventions. The investigators will examine how BA affects early emotional information processing in participants who are currently experiencing low mood, to see whether this can predict eventual changes in mood and to gain a better understanding of the treatment mechanisms of BA. Participants will be in three groups undergoing either behavioural activation, or activity monitoring alone (active control) for 4 weeks, or they will be on a waiting list (passive control). The investigators will also examine whether other factors, such as anxiety, social support and environmental reward, can predict the success of BA. This could help us understand how BA works and who may be most suitable for this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female or male
* Age: 18 to 65 years
* Competency to give informed consent
* Scores above 14 on BDI-2 (bottom criterion for mild depression)

Exclusion Criteria:

* Previous participation in a study that used the emotional test battery (ETB)
* Currently undergoing any form of psychotherapy or counselling
* Taking antidepressant medication for less than 3 months, or changing existing psychiatric medication within the past month
* Current or past a diagnosis of psychosis or a bipolar disorder
* Current diagnosis of an eating disorder, a borderline personality disorder, or a substance abuse disorder
* Any other factor that would indicate the participant isn't able to comply with the requirements of the study according to the opinion of the chief investigator (severe insomnia, chronic fatigue syndrome, neurological conditions impairing cognitive function etc.)
* Symptoms of depression are too severe (score 20 and above on the PHQ-9 questionnaire or according to the evaluation of study psychiatrist)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in recognition of positive and negative facial expressions from baseline at week 2 and 4 | Will be assessed at week 0, week 3 and week 5 of the intervention
  Hit rate for detecting positive versus negative faces in a facial expression recognition task (FERT)

SECONDARY OUTCOMES:
Median scores on the daily Mood Zoom questionnaire | 5 weeks
  Scoring six emotions (Anxious, Elated, Sad, Angry, Irritable and Energetic) on a Likert scale (scale range 1-7). Higher values represent higher levels of the emotion. The six subscales will be combined into 'Positive affect' (Elated, Energetic), 'Negative affect' (Sad, Anxious) and 'Irritability' (Angry, Irritable) scores by averaging.
Motor activity | 5 weeks
  Motor activity (in Hz) as measured by the GeneActive actigraphy watch
Change in speed during recognition of positive and negative facial expressions | Will be assessed at week 0, week 3 and week 5 of the intervention
  Reaction times for correctly recognised positive versus negative faces in facial expression recognition task (FERT)
Change in emotional categorisation (ECAT) | Will be assessed at week 0, week 3 and week 5 of the intervention
  Reaction times for correctly classifying positive versus negative personality characteristic words
Change in recall in the Emotional memory task (EREC) | Will be assessed at week 0, week 3 and week 5 of the intervention
  Number of positive and negative words correctly (and incorrectly) recalled in the EREC task
Change in reward sensitivity | Will be assessed at week 0, week 3 and week 5 of the intervention
  Sensitivity to reward as measured by the Probabilistic Instrumental Learning Task
Change in performance on Auditory Verbal Learning Task (AVLT) | Will be assessed at week 0, week 3 and week 5 of the intervention
  Accuracy on AVLT (number of items recalled across blocks)
Change in levels of behavioural activation | Will be assessed at week 0, week 3 and week 5 of the intervention
  Score on the Behavioural Activation for Depression Scale (total score range 0-150). Higher scores indicate higher levels of activation.
Change in mood | Will be assessed at week 0, week 3 and week 5 of the intervention
  Score on the Beck Depression Inventory (total score range 0-63). Higher scores indicate higher levels of depression.
FERT as a possible predictor of mood change | Will be assessed at week 3 and week 5 of the intervention
  Correlation between Hit rate on the FERT at week 3 and the change in BDI at week 5
Change in environmental reward | Will be assessed at week 0, week 3 and week 5 of the intervention
  Score on the Environmental reward observation scale (total score range 10-40). Higher scores indicate higher levels of environmental reward.
Change in subjective experience of social support | Will be assessed at week 0, week 3 and week 5 of the intervention
  Score on the Multidimensional Scale of Perceived Social Support (total score range 12-84). Higher scores indicate higher levels of support.
Change in anxiety | Will be assessed at week 0, week 3 and week 5 of the intervention
  Score on the State-trait anxiety inventory (both State anxiety and Trait anxiety subscales scores range from 20-80). Higher scores indicate higher levels of anxiety.
EREC as a possible predictor of mood change | Will be assessed at week 3 and week 5 of the intervention
  Correlation between number of correctly recalled positive versus negative personality characteristic words at week 3 and and the change in BDI score at week 5
ECAT as a possible predictor of mood change | Will be assessed at week 3 and week 5 of the intervention
  Correlation between reaction times for correctly classifying positive versus negative personality characteristic words at week 3 and the change in BDI score at week 5
FERT as a possible predictor of mood change | Will be assessed at week 3 and week 5 of the intervention
  Correlation between Reaction times on the FERT at week 3 and the change in BDI at week 5

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided